CLINICAL TRIAL: NCT05339321
Title: A Phase 1 Clinical Study of Autologous HBV-specific TCR-T Cell Therapy (SCG101) in Patients With HBV-related HCC
Brief Title: Autologous HBV-specific T Cell Receptor Engineered T Cells (TCR-T) in Patients With HBV-related Advanced HCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCG101-CI-101
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCG101 (Experimental): SCG101 will be given via Intravenous (IV) infusion.
  Interventions: Genetic: SCG101
- SCG101 + PD1/PD-L1 checkpoint inhibitor (Experimental): SCG101 will be given via Intravenous (IV) infusion. The PD-1/PD-L1 checkpoint inhibitor will be given per product label.
  Interventions: Genetic: SCG101; Biological: PD1/PD-L1 checkpoint inhibitor

INTERVENTIONS:
Genetic: SCG101 — SCG101 is an autologous HBV-specific T cell receptor engineered T cell therapy.
Biological: PD1/PD-L1 checkpoint inhibitor — Commercially approved for HCC treatment.
  Arms: SCG101 + PD1/PD-L1 checkpoint inhibitor

SUMMARY:
Adoptive cell therapy with TCR-T cells targeting HBV antigens represents an innovative opportunity for treatment of HBV-related HCC. SCG101 is a genetically modified autologous TCR-T cell therapy with a natural high-avidity TCR directed towards the HLA-A*02-restricted HBsAg peptide. This is a phase 1 clinical study of SCG101 alone and with PD-1/PD-L1 checkpoint inhibitors in HBV-related HCC.

DETAILED DESCRIPTION:
This is an open-label, multi-center clinical study to evaluate the safety, tolerability and effectiveness of SCG101, with and without PD-1/PD-L1 checkpoint inhibitors, in patients with HBV-related HCC. Lymphodepleting regimen of cyclophosphamide and fludarabine will be given prior to SCG101 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, or imaging diagnosed HCC
2. HLA-A *02 genotyping
3. HBsAg positive in serum or tumor tissue
4. Have at least one measurable lesion at baseline as per mRECIST and RECIST v1.1 criteria
5. Child-Pugh score ≤ 7
6. ECOG performance status of 0 or 1
7. Life expectancy of 3 months or greater
8. Patient with adequate organ function

Exclusion Criteria:

1. Uncontrolled portal vein or inferior vena cava tumor thrombosis
2. Untreated or active Central nervous system (CNS) metastasis or other clinically significant CNS diseases
3. Active or uncontrollable infections
4. History of organ transplantation
5. Lack of peripheral or central venous access or any condition that would interfere with study drug administration or collection of study sample
6. History of positive results for human immunodeficiency virus (HIV) 1 or 2 or known acquired immunodeficiency syndrome (AIDS)
7. Prior exposure to any cell therapy
8. Other severe medical conditions that may limit subject's participation in this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) and laboratory abnormalities defined as dose limiting toxicities (DLT) | 28 days
  To assess the tolerability of SCG101 and determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Efficacy: antitumor activity of SCG101 in subjects with HBV-related HCC | Up to 2 years
  Tumor response assessment in accordance with mRECIST and iRECIST
Efficacy: antiviral activity of SCG101 | Up to 2 years
  Changes in serum levels of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV-DNA) before and after SCG101 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Shunda Du, Principal Investigator — Peking Union Medical College Hospital
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing
  - Zhongshan Hospital, Fudan University, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - The Sixth People's Hospital of Shenyang, Shenyang

REFERENCES:
- [Derived] Wu X, Quan D, Li W, Wisskirchen K, Wu W, Zhou Y, Liu YP, Wan X, Wang X, Zhang X, Yang L, Zheng M, Zhang K, Protzer U, Du S, Qu X. Clinical results of an HBV-specific T-cell receptor-T-cell therapy (SCG101) in patients with HBV-related hepatocellular carcinoma treated in an investigator-initiated, interventional trial. Gut. 2025 Dec 5;75(1):147-160. doi: 10.1136/gutjnl-2025-335456. PMID 40803751
- [Derived] Wan X, Wisskirchen K, Jin T, Yang L, Wang X, Wu X, Liu F, Wu Y, Ma C, Pang Y, Li Q, Zhang K, Protzer U, Du S. Genetically-modified, redirected T cells target hepatitis B surface antigen-positive hepatocytes and hepatocellular carcinoma lesions in a clinical setting. Clin Mol Hepatol. 2024 Oct;30(4):735-755. doi: 10.3350/cmh.2024.0058. Epub 2024 May 29. PMID 38808361